CLINICAL TRIAL: NCT06065800
Title: Assessment of the Performance of STEELEX® Sternum Set + BONE WAX® + STEELEX® Electrode Set in Patients Undergoing Cardiac Surgery. A Prospective, Mono-center, Single-arm, Observational Study in Daily Practice
Brief Title: STEELEX® Sternum Set + BONE WAX® + STEELEX® Electrode Set in Patients Undergoing Cardiac Surgery
Acronym: STEADY
Status: Completed | Type: Observational
Sponsor: Aesculap AG (Industry)
Collaborators: B.Braun Surgical SA (Industry)
Responsible Party: Sponsor
Other Study IDs: AAG-O-H-2045
Record Dates: First submitted 2023-08-24; First posted 2023-10-04 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Sternum Closure
Keywords: non resorbable suture; cardiac surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- STEELEX®: STEELEX® Sternum Set in Patients undergoing cardiac surgery
  Interventions: Device: STEELEX® Sternum Set

INTERVENTIONS:
Device: STEELEX® Sternum Set — Sternal Closure with stainless steel suture (STEELEX®) in patients undergoing cardiac surgery

SUMMARY:
The aim of the study is to assess the effectiveness and performance of using STEELEX® Sternum Set, BONE WAX® and STEELEX® Electrode Set in patients undergoing cardiac surgery. The primary endpoint is the assessment of STEELEX® Sternum Set effectiveness for sternal healing at month 1 ± 1 week post-surgery. This study is designed as a prospective, non-interventional, single center, Post Market Clinical Follow-Up cohort study.

The products under investigation will be used in routine clinical practice and according to the instructions of use. No diagnostic or therapeutic intervention outside of routine clinical practice will be applied, and all study visits will coincide with those that will be scheduled for routine follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients.
* Age ≥ 18 years.
* Scheduled sternotomy within the next 3 days.
* Use of STEELEX® Sternum Set + Bone Wax® for sternotomy following routine clinical practice
* Use of STEELEX® Electrode Set in temporary epicardial cardiac pacing during the postoperative phase of open-heart surgery in combination with an external pacemaker following routine clinical practice.
* Written Informed Consent form.

Exclusion Criteria:

* Participation or planned participation in any clinical trial before study follow-up is completed.
* Pregnancy and/or breastfeeding.
* Patient undergoing emergency surgery.
* Patients taking medical consumption that might affect sternal healing (based on investigator's own clinical criteria)
* Patient with any hypersensitivity or allergy to the components of the medical device.
* Any medical or psychological disorder that, in the investigator's opinion, may interfere with the patient's ability to comply with the study procedures.
* Use of STEELEX® Electrode Set in permanent cardiac pacing or for permanent monitoring.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients undergoing scheduled sternotomy for cardiac surgery
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2023-05-17 (Actual); Primary Completion 2024-11-13 (Actual); Study Completion 2025-04-11 (Actual)

PRIMARY OUTCOMES:
Assessment of STEELEX® Sternum Set effectiveness for sternal healing | at month 1 ± 1 week post-surgery
  The primary variable will be the Sternal Instability Scale (SIS), based on a 4-point scale that is anchored by a grade of 0 that corresponds to a clinically stable sternum with no detectable motion or separation of the sternal edges and a grade 3 that corresponds to a completely separated sternum with marked increased motion or separation of the sternal edges

SECONDARY OUTCOMES:
Assessment of STEELEX® Sternum Set effectiveness for sternal healing | at month 6 ± 1 week post-surgery
  The Sternal Instability Scale (SIS) is a clinical physical assessment tool that aims to assess the stability of the sternum and assign a corresponding grade to the findings of examination. It is based on a 4-point scale that is anchored by a grade of 0 that corresponds to a clinically stable sternum with no detectable motion or separation of the sternal edges and a grade 3 that corresponds to a completely separated sternum with marked increased motion or separation of the sternal edges measured at 6 months postoperative
Rate of sternal dehiscence over time | at month 1 ± 1 week and at month 6 ± 1 week post-surgery.
  Frequency of sternal dehiscence (classified in four types according to the deepness and in two sub-groups according to the vertical extension based on the inferior insertion of the pectoralis major muscle).
Incidence of post-surgery sternal wound complications | at month 1 ± 1 week and at month 6 ± 1 week post-surgery.
  The incidence of post-surgery sternal wound complications at hospital discharge, at month 1 ± 1 week and month 6 ± 1 week post-surgery. Frequency of patients with sternal wound complications at hospital discharge, at month 1 ± 1 week and month 6 ± 1 week post-surgery.
Incidence of post-surgery sternal wound infections | at month 1 ± 1 week and at month 6 ± 1 week post-surgery.
  The incidence of post-surgery wound infections during the 6-month ± 1 week study follow-up. Frequency of wound infections (superficial sternal wound infections [SSWI], or deep sternal wound infections [DSWI]) during the 6-month ± 1 week study follow-up.
Incidence of re-exploration for bleeding over study period | during the first 24-48 hours postoperatively, at hospital discharge (approximately 10 days after surgery), at month 1 ± 1 week
  The incidence of re-exploration for bleeding during the 24-48h post-operation, at hospital discharge and 1-month ± 1 week of study follow-up. Frequency of re-exploration for bleeding until 1-month ± 1 week of study follow-up after surgery.
Incidence of reoperations/readmission after surgery | during the 6-month ± 1 week study follow-up
  The incidence of reoperations/readmission after surgery during the 6-month ± 1 week study follow-up. Frequency of reoperation/readmission after surgery during the 6-month ± 1 week study follow-up.
Length of hospital stay after surgery | at hospital discharge (approximately 10 days after surgery)
  Calculated number of days between surgery and discharge of the patient from hospital
Progress of pain according to the Visual Analogue Scale (VAS) compared to baseline | preoperatively (baseline), at hospital discharge (approximately 10 days after surgery), at month 1 ± 1 week and at month 6 ± 1 week post-surgery.
  The patient's self assessment of pain. This parameter will be noted using the Visual Analogue Scale (VAS), represented by a line 10 cm of length, which states "0" at one end representing "no pain" and "100" at the opposite end representing "heavy pain". The value is measured in [mm] with a ruler and documented in whole numbers.
Rate of adverse device effects (ADEs) | during the 6-month ± 1 week study follow-up.
  The safety profile according to adverse device effects (ADEs) reported after surgery during the 6-month ± 1 week study follow-up. Frequencies of patients with ADEs reported during the 6-month ± 1 week study follow-up after surgery.
Effectiveness of STEELEX® Electrode Set | at hospital discharge (approximately 10 days after surgery)
  The assessment of the STEELEX® Electrode Set effectiveness through the fixation ability of the electrode to the myocardium prior to removal. Percentage of patients with positive or negative myocardial stimulation at hospital discharge.
Mean score of the intraoperative handling questions on STEELEX® Sternum Set and STEELEX® Electrode Set | intraoperatively
  The assessment of the STEELEX® Sternum Set and STEELEX® Electrode Set intraoperative handling through the physician opinion after surgery: Handling of STEELEX® Sternum Set is assessed in five dimensions (on a descending scale from excellent = 5 points to poor = 1 point) in five categories (Knot security, Tensile strength, Needle strength, Passage / Penetration of the needle through the bone, Quality of the connection between the needle and the thread). Handling of STEELEX® Electrode Set is assessed in five dimensions (on a descending scale from excellent = 5 points to poor = 1 point) in four categories (Wire placement in the myocardium, Straight break-off needle connection to the patient cable, Removal of STEELEX® Electrode set of the patient, Tensile strength) The points are added to a handling score ranging from a maximum of 45 to a minimum of 9 points.

CONTACTS AND LOCATIONS:
Overall Officials: Juan Martinez León, Dr., Principal Investigator — Department of Cardiovascular Surgery
Locations (1):
- Department of Cardiovascular Surgery, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No